CLINICAL TRIAL: NCT03477942
Title: A Phase I Single Center Open Study to Assess the Safety and Efficacy of Intra-articular Mesenchymal Stem Cells in the Treatment of Knee Osteoarthritis and Chondral Defects of the Knee
Brief Title: Impact of Mesenchymal Stem Cells in Knee Osteoarthritis
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, James E Voos, MD, Chairman, Department of Orthopaedic Surgery, University Hospitals Cleveland Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY20180044
Record Dates: First submitted 2018-02-22; First posted 2018-03-27 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Musculoskeletal Pain; Knee Osteoarthritis; Cartilage Injury; Cartilage Degeneration
MeSH Terms: conditions — Musculoskeletal Pain; Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Prospective, single-center phase I pilot study to evaluate the safety and tolerability of a single intra-articular injection of autologous bone marrow-derived MSCs in 16 subjects, 8 who have knee osteoarthritis and 8 who have a focal chondral defect in the knee.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Osteoarthritis (Experimental): The OA subgroup will be patients aged 18-60 years who have chronic knee pain due to early OA that have not responded to conservative, non-invasive measures such as physical therapy, medications, and activity modification.
  Interventions: Biological: Autologous Mesenchymal Stem Cells
- Cartilage (Experimental): The focal chondral defect subgroup will be patients aged 18-60 years who participate in recreational or professional sports and are symptomatic from a focal chondral defect shown on MRI.
  Interventions: Biological: Autologous Mesenchymal Stem Cells

INTERVENTIONS:
Biological: Autologous Mesenchymal Stem Cells — Bone marrow will be harvested from each individual patient's iliac crest, followed by stem cell isolation, expansion and preparation. Stem cell will be injected approximately 3-4 weeks after bone marrow harvest, injecting 50x10^6 MSCs in the knee via a medial parapatellar approach under sterile technique in 8 patients with generalized knee OA or focal chondral defects.
  Other Names: Stem Cell Injection

SUMMARY:
Many patients with osteoarthritis of the knee fail non-operative measures and elect to have knee arthroplasty to improve their quality of life. If successful, intra-articular mesenchymal stem cell (MSC) injections into the knee may offer another viable non-operative treatment modality. Additionally, this modality may have reparative or regenerative potential, which could lead to the first treatment for osteoarthritis that treats the underlying disease as opposed to symptomatic control.

Additionally, there are no acceptable non-surgical treatments for focal chondral defects of the knee. Surgical treatments that do exist have diminished outcomes if performed on patients older than age 30-40 years. If successful, intra-articular MSC injections into the knee would represent the first non-operative treatment for focal chondral defects and also represent a potential option for treatment in patients over the age of 30-40 years.

This trial will be a prospective, single-center phase I pilot study to evaluate the safety and tolerability of a single intra-articular injection of autologous bone marrow-derived MSCs in 16 subjects, 8 who have knee osteoarthritis and 8 who have a focal chondral defect in the knee. Patients will undergo a bone marrow harvest procedure at the Dahms Clinical Research Unit (DCRU) of University Hospitals Cleveland Medical Center. MSCs will be isolated and expanded. After approximately 2-3 weeks, patients will return for an intra-articular injection of 50x106 MSCs Subsequent study visits will occur on post-injection day 7 and months 2, 6, 12, and 24. Safety of intra-articular injection of MSCs will be evaluated at study visits by interval history, physical examination and assessment of any adverse events that are observed/reported. Additionally, efficacy will be evaluated by having patients complete functional outcome measures including: Visual Analog Score (VAS) for pain, Knee Injury and Osteoarthritis Outcome Score (KOOS), International Knee Documentation Committee (IKDC) Subjective Knee Form, and Lysholm Knee Scale. These will be completed at the pre-treatment visit and then repeated at the 2, 6, 12, and 24-month follow-up visits. Lastly, T1 rho and T2 mapping on magnetic resonance imaging (MRI) will be used to assess for improved cartilage quality after intra-articular injection of MSCs. An MRI will be obtained at the pre-treatment visit. At the 12 and 24 month follow up visit, additional MRIs will be obtained and analyzed to compare the pre-treatment MRI to post-treatment MRIs.

ELIGIBILITY:
Inclusion Criteria:

Knee Osteoarthritis Subjects

1. Male or female 18-60 years of age
2. Confirmed diagnosis of knee osteoarthritis based on clinical and radiographic findings
3. Unilateral chronic knee pain >4 months
4. Imaging findings consistent with mild-moderate generalized cartilage degeneration (MRI chondropathy or radiographic changes)
5. Failed non-invasive modalities of treatment
6. Subjects must have the ability to understand and the willingness to sign a written informed consent document
7. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use a contraceptive method with a failure rate of <1% per year during the treatment period. A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (<12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). Examples of contraceptive methods with a failure rate of <1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptive that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Period abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception

Focal Chondral Defect Subjects

Inclusion Criteria:

1. Male or female 18-60 year of age
2. Knee pain and/or effusion
3. Inability to continue or difficulty in participation in recreational or professional sport
4. MRI with Outerbridge Grade 4 focal chondral defect
5. Subjects must have the ability to understand and the willingness to sign a written informed consent document
6. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use a contraceptive method with a failure rate of <1% per year during the treatment period. A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (<12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). Examples of contraceptive methods with a failure rate of <1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptive that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Period abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

Exclusion Criteria:

1. Radiographic findings consistent with Kellgren-Lawrence Stage 4 disease
2. Focal chondral defect
3. Major axial deviation (>5 degrees varus or valgus)
4. Concomitant ligamentous or meniscal injury
5. BMI > 40 as defined by NIH Clinical Guidelines Body Mass Index
6. Women who are pregnant, breastfeeding or unwilling to practice birth control during participation in the study
7. Concurrent participation in another investigational trial involving systemic administration of agents (within the previous 30 days), or have received prior intra-articular injection of any form

   • Or plans to participate in any other allogeneic stem cell therapy trial during the 2-year follow-up period
8. Symptomatic active cardiac or respiratory disease that requires scheduled use of medication
9. Neurologic disorder including, but not limited to epilepsy, Parkinson's disease, dementia, cerebrovascular disease, tumor of the nervous system, and amyotrophic lateral sclerosis.
10. Psychiatric disorder including, but not limited to schizophrenia, bipolar disorder, personality disorder, depression, anxiety, or any other mental illness that would prevent the completion of the study
11. Current immunosuppression from medication or disease
12. History of systemic malignancy
13. History of infection with hepatitis B, C, or HIV
14. History of inflammatory arthropathy
15. History of prior local knee infection
16. Major surgeries, other than diagnostic surgery within 4 weeks
17. Contraindication to MRI:

    * Indwelling medical devices such as pacemakers, aneurysm clips, etc.
    * Indwelling metal from any other cause (trauma, etc.). To be excluded with history and/or radiographs, as necessary
18. Screening hematology with white blood cell count < 4.5 x 109 cells/L, hematocrit <30%, and platelets <150 x 109 platelets/L
19. Have a known history of hypersensitivity or anaphylactic reaction to Dimethyl sulfoxide (DMSO)
20. Have been treated in the last 6 months before enrollment for alcohol and/or drug abuse in an inpatient substance abuse program
21. Subject unlikely to complete the study as determined by the Investigator
22. Subjects must have normal marrow function, and be clinically stable with no significant changes in health status within 2 weeks prior to cell collection that the PI/Sub-Investigator deems relevant to exclude from participation. (See below for details of the cell collection procedure)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint: Incidence of treatment emergent major adverse events directly related to MSC injection | 24 months
  Establish the safety and tolerability of expended autologous intraarticular MSC injections into the knee by the incidence of no major adverse events (AE) determined to be directly related to MSC injection by the end of the 24 month follow up period. An AE is any untoward medical occurrence during the clinical investigation in a patient administered stem cells that does not have a causal relationship with the treatment that occurs from the time of consent through the last clinic visit at 24 months post-injection. An AE is therefore any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the administration of the investigational product, whether or not related to that investigational product. AEs will be described by duration (start and stop dates and times), severity, outcome, treatment and relation to investigational product, or if unrelated, the cause.

SECONDARY OUTCOMES:
Secondary Endpoint: Development of Pain following injection based on Visual Analog Scale scoring. | 2, 6, 12 and 24 months
  Pain will be analyzed based on visual analog pain scores (VAS) by clinically and statistically significant amounts by six-month follow up and maintain these improvements throughout the two-year study period. Data analysis will be performed separately on the knee osteoarthritis subgroup and on the focal chondral defect subgroup. This will consist of a comparison of mean values for VAS scoring scales pre-operatively and at follow-up visits at 2, 6, 12, and 24-months. Clinically significant outcomes will be determined based on the minimal clinically important difference (MCID) occurring for each respective scale, which is defined as the smallest change score needed for the effect to be considered clinically relevant; described below. Specifically, VAS represents a patient-reported measurement tool used to quantify perceived level of pain, graded on a scale from 0 to 10 with 0 representing no pain and 10 representing the worse pain possible.
Secondary Endpoint: Clinical Evaluation of Injection based on functional outcomes scoring using KOOS, IKDC and Lysholm scoring scales. | 2, 6, 12 and 24 months
  Functional outcomes will be evaluated clinically and statistically throughout the study period. Data analysis will be performed on the knee osteoarthritis and the focal chondral defect subgroups. Mean values for Knee Injury and Osteoathritis Outcome Score (KOOS), International Knee Documentation Committee Score (IKDC), and Lysholm scoring scales pre-operatively and at follow-up visits at 2, 6, 12, and 24-months will be compared. KOOS is a qualitative assessment of knee pain, stiffness, function, and quality of life within the last week. The IKDC is a quantitative assessment of knee symptoms with daily and sporting activities with a high score of 100 representing no limitations or pain, with lower scores signifying pain or limitations in knee function. The Lysholm score rates knee pain and symptoms with a high score of 100, with scores > 90 representing excellent function and scores <65 representing poor function.
Secondary Endpoint: Reparative potential of intra-articular MSCs based on improvement in cartilage quality using MRI. | 12 and 24 months
  T1 rho and T2 mapping observed from MRIs at 1-year and 2-year follow-up to determine the reparative potential of intra-articular MSCs. T1 rho values increase as degenerative changes worsen; therefore, as cartilage quality improves, it is expected that T1 rho values would increase. T2 mapping values primarily reflect changes in water content and collagen anisotropy. Focal areas of increased T2 mapping values correlate with focal areas of cartilage damage; therefore, as cartilage quality improves, T2 mapping values would decrease. Clinically significant changes will be observed by comparing T1 rho and T2 values in areas of relatively preserved hyaline cartilage within our patients with the areas of degenerative change to utilize an internal control. Data analysis will consist of a comparison of mean values for quantitative T1 rho and T2 mapping data pre-operatively and at follow-up visits at 12 and 24-months.

CONTACTS AND LOCATIONS:
Overall Officials: James E Voos, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospital Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No patient protected health information will be shared outside the primary research team. All patient data will be de-identified.

REFERENCES:
- [Background] Murphy L, Schwartz TA, Helmick CG, Renner JB, Tudor G, Koch G, Dragomir A, Kalsbeek WD, Luta G, Jordan JM. Lifetime risk of symptomatic knee osteoarthritis. Arthritis Rheum. 2008 Sep 15;59(9):1207-13. doi: 10.1002/art.24021. PMID 18759314
- [Background] Sato M, Uchida K, Nakajima H, Miyazaki T, Guerrero AR, Watanabe S, Roberts S, Baba H. Direct transplantation of mesenchymal stem cells into the knee joints of Hartley strain guinea pigs with spontaneous osteoarthritis. Arthritis Res Ther. 2012 Feb 7;14(1):R31. doi: 10.1186/ar3735. PMID 22314040
- [Background] Centeno CJ, Busse D, Kisiday J, Keohan C, Freeman M, Karli D. Increased knee cartilage volume in degenerative joint disease using percutaneously implanted, autologous mesenchymal stem cells. Pain Physician. 2008 May-Jun;11(3):343-53. PMID 18523506
- [Background] Davatchi F, Abdollahi BS, Mohyeddin M, Shahram F, Nikbin B. Mesenchymal stem cell therapy for knee osteoarthritis. Preliminary report of four patients. Int J Rheum Dis. 2011 May;14(2):211-5. doi: 10.1111/j.1756-185X.2011.01599.x. Epub 2011 Mar 4. PMID 21518322
- [Background] Emadedin M, Aghdami N, Taghiyar L, Fazeli R, Moghadasali R, Jahangir S, Farjad R, Baghaban Eslaminejad M. Intra-articular injection of autologous mesenchymal stem cells in six patients with knee osteoarthritis. Arch Iran Med. 2012 Jul;15(7):422-8. PMID 22724879
- [Background] Vega A, Martin-Ferrero MA, Del Canto F, Alberca M, Garcia V, Munar A, Orozco L, Soler R, Fuertes JJ, Huguet M, Sanchez A, Garcia-Sancho J. Treatment of Knee Osteoarthritis With Allogeneic Bone Marrow Mesenchymal Stem Cells: A Randomized Controlled Trial. Transplantation. 2015 Aug;99(8):1681-90. doi: 10.1097/TP.0000000000000678. PMID 25822648
- [Background] Koh YG, Jo SB, Kwon OR, Suh DS, Lee SW, Park SH, Choi YJ. Mesenchymal stem cell injections improve symptoms of knee osteoarthritis. Arthroscopy. 2013 Apr;29(4):748-55. doi: 10.1016/j.arthro.2012.11.017. Epub 2013 Jan 29. PMID 23375182